CLINICAL TRIAL: NCT07140965
Title: The Impact of Surgeon-Interpreted Intraoperative Margin Assessment During Breast Conserving Surgery on Postoperative Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0648; NCI-2025-06199 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-08-21; First posted 2025-08-26 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intraoperative Margin Assessment: Utilizing Intraoperative Margin Assessment during the breast conserving surgery, using pFGS as well as DBT.
  Interventions: Procedure: Pegulicianine Fluorescence-Guided Surgery; Procedure: Digital Breast Tomosynthesis; Procedure: Breast Conserving Therapy

INTERVENTIONS:
Procedure: Pegulicianine Fluorescence-Guided Surgery — Given by Surgery
Procedure: Digital Breast Tomosynthesis — Given by Procedure
Procedure: Breast Conserving Therapy — Given by Procedure

SUMMARY:
To learn if Pegulicianine Fluorescence-Guided Surgery (pFGS), which is part of the Lumicell Direct Visualization System, and Digital Breast Tomosynthesis (DBT) can improve the identification of tumor margins during a partial mastectomy and decrease the need for a second surgery.

DETAILED DESCRIPTION:
Primary Objectives:

-To determine if surgeon interpretation of pFGS and DBT has a higher specificity compared to SEP, resulting in fewer excisions of additional tissue unnecessarily

Secondary Objectives:

* To determine if surgeon evaluation of segmental mastectomy margins using pFGS and DBT is associated with better patient- and physician-reported cosmesis
* To determine if surgeon interpretation of pFGS and DBT results in a lower rate of positive margins after BCS compared to SEP
* To determine if surgeon interpretation of pFGS and DBT has a shorter operative time compared to SEP.
* To determine if surgeon interpretation of pFGS and DBT results in less delays in receipt of adjuvant treatment and the reduction of targeted volume of radiation therapy or omission of radiation altogether

ELIGIBILITY:
Inclusion Criteria:

* We plan to enroll 175 patients.
* Women aged 18 years or older with a breast cancer diagnosis at any stage who will undergo a segmental mastectomy, regardless of receipt of neoadjuvant therapy.

Exclusion Criteria:

1. Multi-site segmental mastectomies within the same breast
2. Participants without a cancer diagnosis
3. Participants from vulnerable populations including minors, pregnant women, and/or cognitively impaired adults.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
safety and adverse events (AEs). Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 6.0 | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Fedra Fallahian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org